CLINICAL TRIAL: NCT04012463
Title: Neural and Behavioral Sequelae of Blast-Related Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Harvey Levin, Professor, Baylor College of Medicine
Other Study IDs: PT074924P1; PT074924P1; H-22852 (Other: Baylor College of Medicine)
Record Dates: First submitted 2015-03-19; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2015-03

CONDITIONS: TBI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis 1: On fMRI scanning, frontoparietal activation during performance of executive function tasks of working memory, inhibitory control processes, and stimulus-response interference will exhibit greater signal intensity, a wider spatial extent, and more bilateral activation in chronic MTBI than chronic OI participants.

Hypothesis 2: DTI changes, characterized by lower FA and higher MD at the gray-white junction, corpus callosum, central semiovale, and internal capsule, will be seen in MTBI but not in OI subjects.

Hypothesis 3: Increased fMRI activation in chronic MTBI will be correlated with location and severity of disrupted fiber tracks that subserve neural networks associated with each fMRI activation task.

Hypothesis 4: Performance on computerized neuropsychological testing (ANAM) and reaction time measures on fMRI tasks will better discriminate MTBI from OI than standard paper-and pencil tests.

Hypothesis 5: The combination of fMRI, DTI, and ANAM will better discriminate MTBI from OI than each individual method.

Hypothesis 6: More severe brain pathology in MTBI, as measured by neuroimaging (fMRI, DTI) and ANAM test scores, will be associated with less severe PTSD and symptoms.

DETAILED DESCRIPTION:
Traumatic brain injuries (TBI) are a common occurrence from roadside blasts of improvised explosive devices (IEDs). Like civilian TBI, blast-related TBI can result from mechanical forces in which objects in motion strike the head or the head is forcefully put into motion and strikes an object. TBI from exposure to an explosive blast may also result from a third cause: barotrauma. Blasts produce wave-induced changes in atmospheric pressure, which in turn produce characteristic injuries to vulnerable bodily regions at air-fluid interfaces, such as the middle ear. It is unknown whether the neural and cognitive sequelae of blast-related TBI differ from those resulting from mechanically-induced TBI commonly observed in civilian accidents. Understanding the potentially unique sequelae of blast-related TBI is critical for accurate diagnosis and designing effective pharamacological and neurorehabilitation interventions.

In the proposed cross-sectional study, we aim to apply neurobehavioral testing and advanced MRI techniques [task-activated functional MRI (fMRI) and diffusion tensor imaging (DTI)] to gain a comprehensive understanding of the neural changes underlying blast-related MTBI. This will be accomplished by comparing neurobehavioral and neuroimaging findings obtained from military personnel who have experienced a blast injury with those obtained from civilians who have experienced TBI from motor vehicle accidents and from military and civilian control participants with orthopedic injuries. We will accomplish this goal by conducting advanced neuroimaging (task-activated fMRI and DTI fiber tracking) and neurobehavioral testing (computerized assessment and standard neuropsychological testing) on 120 chronic trauma patients: 30 military MTBI patients who have experienced blast injuries, 30 civilian MTBI patients with mechanical closed head injuries, and 30 military and 30 civilian patients with orthopedic injuries.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for milMTBI

1. GCS score 9-15 (if available) 2. Brain injury due to blast 3. Current age 18-45 4. Right-handed 5. Post-injury interval 12-72 months 6. Duration of Loss of Consciousness (LOC) < 24 hours 7. Duration of Posttraumatic Amnesia (PTA)< 7 days 8. No intracranial surgery 9. No brain lesions on computer tomography (CT) scan (if available) 10. Extracranial Injuries by Abbreviated Injury Scale (AIS) <3 (non-head)

Inclusion Criteria for civlMTBI

1. GCS score 9-15 (if available) 2. Non-blast brain injury 3. Current age 18-45 4. Right-handed 5. Post-injury interval 12-72 months 6. LOC < 24 hours 7. PTA< 7 days 8. No intracranial surgery 9. No brain lesions on CT scan (if available) 10. Extracranial Injuries by AIS <3 (non-head)

Inclusion Criteria for milControl and civOI

1. No history of brain injury 2. Non-blast extracranial injury or no injury 3. Current age 18-45 4. Right-handed 5. Post-injury interval 12-72 months 6. LOC -none 7. PTA- none 8. No intracranial surgery 9. CT scan normal (if done) 10. Extracranial Injuries by AIS <3 (non-head)

Exclusion Criteria:

1) Not fluent in English 2) Non-right hande 3) AIS score equal or higher 4 for body parts other than head 4) Neurologic deficit other than TBI (MTBI, OI groups); no LOC or PTA (MTBI groups) 5) Blood alcohol level > 200 mg/dL 6) Previous hospitalization for head injury 7) Pregnancy when screened prior to brain imaging 8) Pre-existing neurologic disorder associated with cerebral dysfunction and/or cognitive deficit (e.g., cerebral palsy, mental retardation, epilepsy) or diagnosed dyslexia 9) Pre-existing severe psychiatric disorder (bipolar disorder, schizophrenia) as determined by the Structured Clinical Interview for Depression 10) Penetrating gunshot wound to the brain 11) Contraindications to undergoing MRI, including implant of metal or marked agitation observed by research assistant. 12) Illegal alien 13) Hypoxia for 30 minutes or longer after resuscitation PO2 < 96 mmHg 14) Hypotension for 30 minutes or longer after resuscitation (systolic blood pressure more than 2SDs below mean for age)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a prospective, observational study using a cross-sectional design to compare brain imaging and neuropsychological findings at 12 to 72 months post-injury in four groups of at least 30 patients each: two groups of military patients who have sustained mild to moderate TBI (milMTBI) or orthopedic injury or uninjured veterans, reservists, or service members (milControl) and two groups of civilian patients who had MTBI (civMTBI) or OI (civOI).
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Brain activation on Stop Signal Reaction Time Task (SSRT) | 12-24 months post-injury
  fMRI measuring brain activation associated with performance of SSRT
Brain activation on Sternberg Item Recognition Task (SIRT) | 12-24 months post-injury
  fMRI measuring brain activation associated with performance of SIRT

SECONDARY OUTCOMES:
Neurobehavioral Symptom Inventory | 12-24 months post-injury
  self-report of various domains of emotional status
Post-traumatic Symptom Checklist-Civilian (PCL-C) | 12-24 months post-injury
  Checklist of posttraumatic stress symptoms
Center for the Epidemiological Center for Study of Depression (CES-D) | 12-24 months post-injury
  Self-report measure of depression
Symbol Digit Modalities Test (SDMT) | 12-24 months post-injury
  Measure of processing speed
Trail Making Test A and B | 12-24 months post-injury
  Measure of visuoperceptive performance and speed
Controlled Oral Word Association | 12-24 months post-injury
  Measure of verbal fluency
California Verbal Learning Test 2 | 12-24 months post-injury
  Verbal learning test

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Levin, PhD, Principal Investigator — Baylor College of Medicine; Steven Rao, PhD, Principal Investigator — The Cleveland Clinic